CLINICAL TRIAL: NCT05549375
Title: Neurorehabilitation of the Hand
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IRegained Inc. (Industry)
Collaborators: Laurentian University (Other); Health Sciences North (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LUSUON0001
Record Dates: First submitted 2021-07-28; First posted 2022-09-22 (Actual); Last update posted 2022-09-22 (Actual); Status verified 2022-09

CONDITIONS: Stroke
Keywords: Hand Function; Rehabilitation; Engagement; Motor control
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Neurorehabilitation of the Hand (Experimental)
  Interventions: Device: MyHand System Hand Rehabilitation

INTERVENTIONS:
Device: MyHand System Hand Rehabilitation — 15 1-hour patient specific sessions using the MyHand System to help improve Hand function in the affected hand of stroke survivors

SUMMARY:
Stroke is the number one cause of adult disability in the world. Due to the neurological damage from stroke, a vast majority of individuals suffer from hand function disability (~70%). To improve hand function and overcome challenges from this disability, IRegained has developed the MyHandTM system, a connected mechatronic device with programmed proprietary hand function training protocols developed through deep research in neuroplasticity that provide targeted hand function therapy. When these therapeutic protocols are provided in a gamified format, it enhances the patient engagement and motivation, thereby enabling effective therapy administration with the required intensity and repetition to improve hand function. Participants who have sustained a stroke 6 months or earlier will be eligible to participate in this study, and will undergo hand function therapy for one 1-hour/session, 5 times/week, over a 3-week duration, for a total of 15 sessions. Therapy will be administered through with specific hand functions in a gamified format to enhance greater function in the hand and thereby help patients gain greater independence in performing activities of daily living. This research project will aim to understand the extent to which this approach to therapy impacts patient motivation and engagement in order to develop the most efficient and effective mode of therapy.

ELIGIBILITY:
Inclusion Criteria:

* sustained a single stroke
* aged between 30-85 years of age.

Exclusion Criteria:

* Participants with severe spasticity or contractures,
* have other musculoskeletal or neuromuscular disorders that compromises sensation or other neuromuscular parameters
* participants who are unable to provide consent to participate

Ages: 30 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2021-08-04 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
the Nasa-Task Load Index (NASA-TLX) | immediately after each treatment session
  an assessment tool used to evaluate the participant's perceived cognitive load during an activity will be used. It has six subscales; mental demand, physical demand, temporal demand, performance, effort, and frustration. To estimate the level of participant engagement, the participants score within the game/intervention, the time taken to complete a level, as well as verbal language references made during gameplay will be utilized along with the NASA-TLX sub-scores
ABILHAND- change is being assessed | Baseline- prior to intervention and post- intervention- one day after completing the intervention
  ABILHAND a subjective functional assessment tool will be used. The tool is a 23-item survey, and participants are provided with a list of various everyday functional tasks and are scored based on patient response. For example, participant will be asked whether it is 'easy', 'difficult' or 'impossible' for each of the 23 tasks.
Jebson Taylor Hand Function Assessment-change is being assessed | Baseline- prior to intervention and post- intervention- one day after completing the intervention
  7 tasks used to measure participants functional ability with they upper limbs

CONTACTS AND LOCATIONS:
Overall Officials: Ratvinder Grewal, Principal Investigator — Laurentian University
Locations (1):
- Norcat, Greater Sudbury, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided